CLINICAL TRIAL: NCT04761653
Title: Prognostic Impact of the Inflammatory Microenvironment in Atypical Meningiomas
Brief Title: Study of the Inflammatory Microenvironment in Atypical Meningiomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Guillaume GAUCHOTTE, PU PH, Central Hospital, Nancy, France
Other Study IDs: 2021PI015
Record Dates: First submitted 2021-02-16; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Atypical Meningioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — FFPE tissue block
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atypical meningiomas represent 15% of meningiomas. They present a high rate of recurrence, and therapeutic strategies are limited. There is a need for novel treatment strategies, such as immuotherapy.

This is a retrospective study including 84 patients with primary diagnosis of atypical meningiomas. The presence of T cells (CD4, CD8, Treg and memory T cells) and mature dendritic cells will be quantified on whole tissue sections stained by immunohistochemistry (CD4, CD8, FOXP3, CD45RO and CD208).

This could allow us to identify novel biomarkers for survival, and facilitate the selection of patients who may benefit from immunotherapeutic modalities.

ELIGIBILITY:
Inclusion Criteria:

* primary diagnosis of atypical meningioma
* surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated for a cerebral tumor, with primary diagnosis of atypical meningioma
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2-21 years

SECONDARY OUTCOMES:
Overall survival | 2-21 years

CONTACTS AND LOCATIONS:
Locations (1):
- Guillaume GAUCHOTTE, Vandœuvre-lès-Nancy, France